CLINICAL TRIAL: NCT00244075
Title: Effects of Nutritional Supplementation on Protein and Energy Homeostasis in Malnourished Chronic Hemodialysis Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Alp Ikizler, Professor, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9458
Record Dates: First submitted 2005-10-21; First posted 2005-10-25 (Estimated); Last update posted 2015-05-25 (Estimated); Status verified 2015-05

CONDITIONS: End Stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Dietary Supplements; Growth Hormone; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): nutrition supplementation, recombinant human growth hormone, and exercise
  Interventions: Dietary Supplement: nutritional supplement; Drug: recombinant human growth hormone (rcGH); Behavioral: exercise
- 2 (Active Comparator): nutrition supplementation only
  Interventions: Dietary Supplement: nutritional supplement

INTERVENTIONS:
Dietary Supplement: nutritional supplement — either oral nutritional formula (Nepro) or intravenous IDPN solution will be administered during hemodialysis; Nepro has a total calorie amount as well as protein, carbohydrate and fat content that are comparable to that of IDPN, and will be provided at four equal amounts with 1-hour intervals throughout the study (150 ml for a total of 600 ml over 4 hours of hemodialysis); IDPN consists of 225 ml of amino acids at a concentration of 15%, 112.5 ml of dextrose at 50% and 112.5 ml of lipids at 20%, will be given at a rate of 150 ml/hr, and will provide 209 kcal/hr
Drug: recombinant human growth hormone (rcGH) — subcutaneous administration of 75 micrograms/kg/day of rcGH for 3 consecutive days
  Arms: 1
Behavioral: exercise — either dual leg press (3 sets of 8-12 repetitions) beginning 30 minutes prior to hemodialysis, or modified stepper (minimum of 15 minutes up to a maximum of 90 minutes, depending upon the patient's tolerance) beginning 15 minutes post initiation of hemodialysis
  Arms: 1

SUMMARY:
The goal of this study is to evaluate the metabolic effects of concomitant use of three consecutive doses of recombinant human growth hormone over three days and exercise during continuous nutrient infusion in chronic hemodialysis patients. We would also like to evaluate the metabolic effects of nutritional supplementation alone without the additional anabolic strategies.

ELIGIBILITY:
Inclusion Criteria:

* On hemodialysis for more than 6 months, on a thrice weekly hemodialysis program;
* Adequately dialyzed (Kt/V > 1.4).

Exclusion Criteria:

* Patients unable to perform exercise.
* Pregnant women.
* Severe unstable underlying disease besides commonly associated with ESRD. Cardiac patients that are stable will be included.
* Patients hospitalized within the last month prior to the study.
* Patients with recirculation detected on the AV graft.
* Patients receiving steroids and/or other immunosuppressive agents

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 1998-07; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
net muscle protein balance | 10 hours

SECONDARY OUTCOMES:
net whole body protein balance | 10 hours

CONTACTS AND LOCATIONS:
Overall Officials: Alp Ikizler, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States

REFERENCES:
- [Result] Pupim LB, Flakoll PJ, Ikizler TA. Nutritional supplementation acutely increases albumin fractional synthetic rate in chronic hemodialysis patients. J Am Soc Nephrol. 2004 Jul;15(7):1920-6. doi: 10.1097/01.asn.0000128969.86268.c0. PMID 15213282
- [Result] Ikizler TA, Pupim LB, Brouillette JR, Levenhagen DK, Farmer K, Hakim RM, Flakoll PJ. Hemodialysis stimulates muscle and whole body protein loss and alters substrate oxidation. Am J Physiol Endocrinol Metab. 2002 Jan;282(1):E107-16. doi: 10.1152/ajpendo.2002.282.1.E107. PMID 11739090
- [Result] Pupim LB, Flakoll PJ, Levenhagen DK, Ikizler TA. Exercise augments the acute anabolic effects of intradialytic parenteral nutrition in chronic hemodialysis patients. Am J Physiol Endocrinol Metab. 2004 Apr;286(4):E589-97. doi: 10.1152/ajpendo.00384.2003. Epub 2003 Dec 16. PMID 14678952
- [Derived] Mah JY, Choy SW, Roberts MA, Desai AM, Corken M, Gwini SM, McMahon LP. Oral protein-based supplements versus placebo or no treatment for people with chronic kidney disease requiring dialysis. Cochrane Database Syst Rev. 2020 May 11;5(5):CD012616. doi: 10.1002/14651858.CD012616.pub2. PMID 32390133